CLINICAL TRIAL: NCT06711666
Title: Prenatal Maternal Mental Health and Neurodevelopment in Children With an Antenatal Diagnosis of Congenital Heart Disease: The Neuro-Moms CHD Study
Brief Title: Prenatal Maternal Mental Health and Neurodevelopment in Congenital Heart Disease
Acronym: Neuro-Moms
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C23-22; 2024-A02138-39 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-11-20; First posted 2024-12-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Congenital Heart Disease; Cyanotic Congenital Heart Disease; d-Transposition of the Great Arteries; Hypoplastic Left Heart Syndrome
Keywords: psychological stress; Maternal prenatal mental health; Neurodevelopment; Cyanotic congenital heart disease; Prenatal diagnosis
MeSH Terms: conditions — Heart Defects, Congenital; Hypoplastic Left Heart Syndrome; Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital heart disease (CHD) is the leading cause of congenital malformations, representing 1% of live births. Progress in surgical care have led to the dramatic increase in the population of children and adults living with heart disease. As survival is no longer a concern, long-term outcomes have become the major public health issue. Prenatal diagnosis of CHD requiring open-heart surgery can be a traumatic event for expecting mothers and fathers. In the general population, maternal mental health distress is associated with fetal disturbances in the hypothalamic-adrenal-pituitary system axis, restricted intrauterine growth and adverse outcomes in the offspring. It is unknown whether prenatal maternal psychological distress have an impact on neurodevelopmental outcomes in CHD. Our national study seeks to (1) characterize the impact of prenatal maternal psychological distress on neurodevelopmental outcomes at age 1 for children with CHD who undergo neonatal open-heart surgery; (2) investigate the sociodemographic and medical determinants associated with prenatal maternal mental health of women carrying a foetus diagnosed with complex CHD; (3) explore the mediating role of prenatal risk factors (i.e., sociodemographic, medical and maternal coping mechanisms) in the association of prenatal maternal mental health (i.e., distress, anxiety and depression) and neurodevelopment in children with CHD; and (4) explore the impact of paternal or the co-parent's mental health impact on neurodevelopmental outcomes at age 1 in children with CHD. This study is a non-interventional, prospective, and longitudinal study of prenatal maternal mental health and subsequent child's neurodevelopmental and behavioural outcomes. It includes a follow-up period from the 3rd trimester of pregnancy until the child's first year of life. It will include children with a prenatally diagnosed heart defect requiring open-heart surgery within the first weeks of life. Understanding and preventing the neurodevelopmental sequelae of heart disease diagnosed in-utero is a public health priority.

DETAILED DESCRIPTION:
This study is a non-interventional, prospective, and longitudinal study of prenatal maternal mental health and subsequent child's neurodevelopmental and behavioural outcomes in congenital heart disease. It includes a follow-up period from the 3rd trimester of pregnancy until the child's first year of life (between 12 and 18 months). It will include children with a prenatally diagnosed critical heart defect (i.e., cyanotic types of CHD with the potential to cause rapid hypoxemia after birth) requiring neonatal open-heart surgery (within the first weeks of life).

Expecting mothers who agree to participate will undergo comprehensive psychological evaluations conducted by a licensed mental health professional with defined expertise in perinatal mental health. Fathers or co-parent of the child with foetal CHD will also participate in self-reports during the prenatal period. A total of three time points of psychological assessment will be done: Time 1, during the prenatal period, after 28 weeks of gestation); Time 2, an interim self-report assessment using only questionnaires before post-surgery hospital discharge for the baby (after intensive care transfer to hospitalization); and Time 3, 1 year after the birth of their child. Maternal assessments will include standardized self-report measures of stress, anxiety, depression and other psychological symptoms as well as a clinical interview for Time 1 and 2. Co-parent assessment at Time 1 will include self-reports of overall mental health, anxiety and coping skills.

Infant neurodevelopmental and behavioural assessments will be conducted at year 1 (between 12-18 months for the child) during a joint visit of the dyad mother-child. All assessments will be standardized and have French norms and instructions for parents and the child. These assessments will evaluate areas such as cognition, emerging language, and motor skills (gross and fine motor abilities). Socio-behavioural outcomes will also be evaluated at this time. All infant developmental assessments will be administered by paediatric neuropsychologists.

ELIGIBILITY:
Inclusion Criteria for the mother of a child diagnosed with CHD:

1. Age at least 18 years old
2. Expecting women
3. Having received a diagnosis of foetal critical cyanotic CHD (i.e., CHD physiology that can compromise blood oxygenation after birth). This type of CHDs corresponds to the highest level of neurological risk as reported by the American Heart Association guidelines(1).
4. Pregnancy of at least 28 weeks of gestation (third trimester) and up to the 38 weeks of gestation at the time of enrolment and prenatal visit for the study.
5. Medical maternal and paediatric cardiology follow-up in one of the investigating hospitals (Montpellier, Necker Children's Hospital in Paris and Bordeaux).
6. A delay of a minimum of 4 weeks between the initial diagnosis of foetal congenital heart disease.
7. Social security affiliation in France.

Inclusion criteria for the father or co-parent:

1. Co-parent of an expecting woman participating in the study
2. Age at least 18 years old
3. Social security affiliation in France.

Inclusion criteria for the child diagnosed with congenital heart disease:

1. Child with a prenatal diagnosis of isolated complex congenital heart disease, born to a mother already participating in the study
2. Written consent from both parents
3. Social security affiliation in France.

Exclusion Criteria for mothers:

1. Patient refusal to participate
2. Participants (i.e., expecting women) who express a wish for medical termination of pregnancy
3. Diagnosis of a complex CHD associated with another foetal comorbidity with a clinically recognized impact on neurodevelopment (e.g., genetic syndromes such as trisomies, poly-malformation syndromes).
4. Participants who are not able to understand the instructions and/or complete the self-reports
5. Expecting women who currently have a major psychiatric condition (e.g., untreated major depression, severe anxiety disorders, psychotic disorders) with or without treatment, at the time of the cardiology consultation or at the time of the first psychological evaluation. Patients who will be excluded due to these conditions will be referred for perinatal psychiatric consultation.
6. Persons under legal or judicial guardianship.

Exclusion Criteria for fathers or co-parents:

1. Patient refusal to participate
2. Participants with a severe psychiatric disorder (severe depression, psychotic disorders) with or without treatment
3. Persons under legal or judicial guardianship.

Exclusion Criteria for children with CHD:

1. Genetic anomalies, brain malformations that may render difficult the neurodevelopmental assessment.

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Expecting women diagnosed with a foetal complex congenital heart disease. Fathers or co-parent of prenatally diagnosed children with CHD Children with complex congenital heart disease who require neonatal open-heart surgery.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Global Mental Health Self-questionnaire, The Symptom Checklist-90-Revised SCL-90 R (min score 20 - max score 80) | Time 1 Prenatal Visit and Time 3 1-year old Visit
  Mental Health Self-Report, Higher scores indicate worse outcomes
Bayley Scales of Infant and Toddler Development (BAYLEY-4) (min score 50- max score 150) | Time 3 1-year old Visit
  Standardized Neurodevelopmental Assessment, Higher scores better outcome, Mean 100; SD 15

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI-Y) (min score 20 - max score 80) | Time 1 Prenatal Visit, Time 2 immediately after the neonatal open-heart surgery during postoperative hospitalization, Postoperative Visit and Time 3 1-year old Visit
  Anxiety self-report, Higher scores worse outcomes
Coping Inventory for Stressful Situations (CISS), (min score 20 - max score 80) | Time 1 Prenatal Visit and Time 3 1-year old Visit
  Coping self-report, Higher scores better outcomes
Post-partum depression Edinburgh Scale (EPDS) (min score 0 - max score 30) | Time 2 immediately after the neonatal open-heart surgery during postoperative hospitalization, Postoperative Visit
  Post-partum depression self-report, Higher scores worse outcomes
Post-Traumatic Stress Scale (PCL-5), (min score 0 - max score 80) | Time 3 1-year old Visit
  Self-report scale on PTSD symptoms, Higher scores worse outcomes
Ages and Stages Parent Report, 3rd Edition (min score 0 - max score 60) | Time 3 1-year old Visit
  Developmental questionnaire for parents, Higher scores worse outcomes

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Hopital de Marseille la Timone, Marseille
  - CHU de Montpellier, Montpellier
  - Institut Saint Pierre, Palavas-les-Flots
  - Hopital Necker Enfants Malades, Paris
  - Hopital Haut Leveque, Pessac

REFERENCES:
- [Derived] Deninotti J, Derridj N, Martins S, Laux D, Stos B, Levy M, Desnous B, Guillaumont S, Amedro P, Chabaneix J, Pfister M, Marguin G, Desmure G, Vincenti M, Bonnet D, Calderon J. Prenatal maternal mental health and neurodevelopment in congenital heart disease in France: the neuro-moms CHD multicentre prospective study protocol. BMJ Open. 2025 Dec 23;15(12):e104889. doi: 10.1136/bmjopen-2025-104889. PMID 41436266
- See also: Video Neuro-Moms CHD — https://www.youtube.com/watch?v=Iph2s9J08sQ